CLINICAL TRIAL: NCT07069192
Title: The Effect of Passive Smoke Exposure and Counselling Intervention in Childhood Asthma
Brief Title: The Invisible Trigger: A Quasi-Experimental Study on the Effect of Passive Smoke Exposure and Counselling Intervention in Childhood Asthma
Acronym: Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Principal Investigator, Ayesha Saeed, Public health Officer, Foundation University Islamabad
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FUMCRCT1
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Childhood Asthma; Passive Smoke Exposure
Keywords: Asthma.; Passive Smoke Exposure,; Secondhand Smoke,; Counsel Intervention,; Childhood Asthma,; Asthma Control Test,; Caregiver Education
MeSH Terms: conditions — Asthma | interventions — Counseling

STUDY DESIGN:
Intervention Model Description: The primary purpose is to offer practical insights into reducing the burden of childhood asthma by fusing exposure reduction techniques with asthma management education. It is anticipated that the results will guide evidence-based policy and public health campaigns to lower exposure to SHS, improve asthma outcomes, and improve the lives of children with the condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): usual care without counselling
- Counselling (Experimental): Counselling
  Interventions: Behavioral: Counselling

INTERVENTIONS:
Behavioral: Counselling — Received structured caregiver counseling - weekly sessions for 1 month and biweekly for the next 2 months.
  Arms: Counselling

SUMMARY:
This study evaluates the effect of passive smoke exposure on childhood asthma and the role of structured counseling in reducing SHS exposure and improving asthma control.

DETAILED DESCRIPTION:
A quasi-experimental study conducted at Fauji Foundation Hospital using a pre-post test design. The intervention group received structured caregiver counseling about the dangers of passive smoking and asthma management. The study used ACT scores to assess improvement in asthma control.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Asthma, Passive smoke exposure

Exclusion Criteria:

* Comorbidity, sever asthma requiring hospitalisation

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 126 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Asthma control test (ACT) Score Improvement | 3 months
  Change in ACT Score from baseline to 3 months after intervention. ACT score of 19 is considered as normal Asthma control, less then 19 is considered as poor Asthma control and more than 19 ACT score is considered as good Asthma control

CONTACTS AND LOCATIONS:
Locations (1):
- Fauji Foundation Hospital, Rawalpindi, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Not Required